CLINICAL TRIAL: NCT07151469
Title: Kaltenborn Mobilization Versus Active Release Technique on Temporomandibular Joint Dysfunction for Radiation - Induced Trismus in Patients With Head and Neck Cancer
Brief Title: Kaltenborn Versus Active Release on Temporomandibular Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005945
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kaltenborn mobilization (Experimental): A certified therapist administered TMJ KM in the following way. The therapist stood behind the seated patient, placing their palms on both sides of the patient's head, with the thumbs over the zygomatic arches, to stabilize the head.
  Interventions: Other: Kaltenborn mobilization
- active release technique (Experimental): This deep tissue therapy technique is primarily used to break up adhesions and scar tissue on the surrounding muscle and ligaments. However, this technique has been proven to be a very effective method for treating TMD
  Interventions: Other: active release technique
- control (No Intervention): No intervention

INTERVENTIONS:
Other: Kaltenborn mobilization — The therapist applies gentle traction to the mandible, maintained for approximately 20 to 30 seconds, to create space in the joint. This is done by pulling the jaw downward and slightly forward, which can help alleviate pressure and pain. This hand placement allowed the therapist to apply transverse force across the mandible as necessary, while at the same time allowing an anterior-inferior gliding force to the mandible on the side of restriction, while also controlling the unrestricted side inhibiting any excessive mandibular forward gliding with the other hand. The mobilization is then initiated with Grade I, which involves small-amplitude movements performed at the beginning of the range of joint play to reduce pain and muscle guarding. This is followed by Grade II mobilization, which consists of larger amplitude movements within the mid-range of joint play to enhance joint mobility and decrease pain without reaching the joint's full resistance barrier
  Arms: Kaltenborn mobilization
Other: active release technique — This deep tissue therapy technique is primarily used to break up adhesions and scar tissue on the surrounding muscle and ligaments. However, this technique has been proven to be a very effective method for treating TMD.While there are several muscles connected with the movement of the TMJ, it is thought that the major players are the digastricus, masseter, and lateral pterygoid muscles
  Arms: active release technique

SUMMARY:
Temporomandibular disorder (TMD) is a term describing musculoskeletal conditions of the face, jaw and temporal regions. TMD is frequently associated with pain and/or dysfunction such as impaired jaw function, pain in the temporomandibular joint (TMJ), muscles and/or related structures, and associated headaches. The etiology of TMD is multifactorial and complex.

It is known that one cause of TMD symptom development is treatment for head and neck cancer (HNC). The main treatment modalities for HNC include radiotherapy (RT) with or without chemotherapy and surgical intervention, as either a single therapy or a combination therapy. In the head and neck region, the anatomical structures are necessary for essential functions such as speech, swallowing, breathing, smell, and taste. The treatment of head and neck tumors may frequently impair some of these functions, which may result in pain, oral dysfunction, and impaired health-related quality of life.

DETAILED DESCRIPTION:
KMT evaluates the motions on the articular surfaces and applies them to treatment according to MacConaill's classification of synovial joints to restore the reduced accessory glides and achieve painless physiological movements. KMT involves the application of a passive sustained joint play that can be graded from I to III based on the type and amount of force applied. Grade-I, "loosening" refers to small-amplitude joint distraction that produces an appreciable increase in joint separation without any stress on the capsule that equalizes the cohesive forces, muscle tension and atmospheric pressure acting on the joint. Grade-II, "tightening" refers to the distraction or glide movements applied to tighten the tissues around the joint, also known as "taking up the slack". Grade-III, "stretching" refers to the distraction or glide movement applied to stretch the joint capsule and surrounding per articular structures, thus, increasing joint ROM.

Another option to consider is offered here at Pain and Performance Solutions. We have seen great results from treating TMJ disorders using Active Release Technique®. This deep tissue therapy technique is primarily used to break up adhesions and scar tissue on the surrounding muscle and ligaments. However, this technique has been proven a very effective method for treating TMD.

ELIGIBILITY:
Inclusion Criteria:

* An experienced oral and maxillofacial surgeon will diagnose patients with temporomandibular joint disorders (myofascial pain, trismus and limitation of ROM) after head and neck cancer, patients.
* Patients with 20 to 60 years old.
* 6 months after ending radiotherapy.

Exclusion Criteria:

* Patients with implants.
* Current metastasis.
* Continuing radiotherapy.
* Pregnant females.
* Sensitivity to phototherapy.
* Bell's palsy.
* Subjects with disk displacement, arthralgia or osteoarthritis at TMJ.
* Subjects who received analgesics or antidepressants.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-02-10 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | at baseline and at 8 weeks
  The pain pressure threshold over the temporalis and masseter muscles will be assessed using an algometry with a 1 cm2 probe tip.lower thresholds indicating increased tenderness and sensitivity
Maximal interincisal opening | at baseline and at 8 weeks
  The stainless steel vernier caliper, which has two arms-one fixed and one movable-connected by a calibrated scale, showed exceptional reliability for measuring mouth opening.Millimeters were used to measure the separation between the incisal edges of the upper and lower incisor teeth

SECONDARY OUTCOMES:
Functional disability | at baseline and at 8 weeks
  It will be measured by jaw functional limitation scale-20. It has a score range of 1 to 200, and high scores indicate worsening jaw function.
Quality of life (Oral health Impact Profile | at baseline and at 8 weeks
  By using the Oral health, Impact Profile consisted of 7 different domains (functional limitation, physical pain, psychological discomfort, psychological disability, physical disability, social disability, and handicap).a 5-point Likert scale (zero = never to four = very often). A summing of the domain scores derived the total score; it can range from zero to 56. A higher score indicates a poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt